CLINICAL TRIAL: NCT01513135
Title: A Phase Il, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Immunogenicity and Safety of a Therapeutic, Recombinant, Biologically Active HIV-1 Tat Protein Vaccine in HIV-Infected, Anti-Tat Negative, ARV-Treated Adult Volunteers
Brief Title: A Phase Il of a Therapeutic, Recombinant, Biologically Active HIV-1 Tat Protein Vaccine in HIV-Infected, Anti-Tat Negative, ARV-Treated Adult Volunteers
Acronym: ISS T-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ensoli, MD (Other)
Collaborators: Italian Ministry of Foreign Affairs - General Direction for Cooperation and Development (Unknown)
Responsible Party: Sponsor-Investigator, Barbara Ensoli, MD, PhD, Istituto Superiore di Sanità
Organization: Istituto Superiore di Sanità (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISS T-003
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infections
Keywords: HIV,; HAART-treated; participants; Tat protein,; Therapeutic immunization
MeSH Terms: conditions — HIV Infections | interventions — tat Gene Products, Human Immunodeficiency Virus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A, Tat (Experimental): Recombinant biologically active Tat 30 mcg in Phosphate saline buffer, pH 7.4, 1% sucrose, 1% Human Serum Albumin; administered intradermally 3 times at weeks 0, 4 & 8
  Interventions: Biological: Tat
- group B, Placebo (Placebo Comparator): Phosphate saline buffer, pH 7.4, 1% sucrose, 1% Human Serum Albumin, administered intradermally 3 times at weeks 0, 4 & 8
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Tat — Recombinant biologically active Tat 30 mcg in Phosphate saline buffer, pH 7.4, 1% sucrose, 1% Human Serum Albumin
  Arms: Group A, Tat
Biological: Placebo — Phosphate saline buffer, pH 7.4, 1% sucrose, 1% Human Serum Albumin
  Arms: group B, Placebo

SUMMARY:
Tat is a key HIV regulatory protein produced very early after infection, prior to virus integration, and necessary for viral gene expression, cell-to-cell virus transmission and disease progression. Previous studies in natural HIV infection, indicated that the presence of a Tat-specific immune response correlates with a lower incidence and reduced risk of progression to AIDS as compared to anti-Tat negative individuals suggesting that an immune response to Tat may exert a protective role and control the progression to AIDS in vivo. Moreover, Tat is conserved in its immunogenic regions (both B and T cell) among all subtypes. subtypes. Recent data, in fact, indicate an effective cross-clade recognition of clade B strain-derived (BH-10) Tat protein from the HTLV-IIIB lab-adapted virus strain (Buttò, 2003), which was isolated about 30 years ago (Ratner, 1985), by sera from individuals infected with viruses circulating at the present in Italy and in Africa, thus reflecting the high degree of conservation of the corresponding Tat regions and providing strong formal evidence that a Tat-based vaccine may indeed be used in the different geographic areas of the world, since it is capable of inducing a broad immune response against different virus clades. Based on this rationale and on the positive results of preclinical (Cafaro, Nat Med 1999) and phase I preventive and therapeutic clinical trials with Tat protein (ISS P-001 and ISS T-001, respectively) (Ensoli AIDS 2008, Vaccine 2009; Longo Vaccine 2009; Bellino RRCT, 2009) a phase II therapeutic, open label, clinical study with Tat protein (ISS T-002, ClinicalTrials.gov NCT00751595) was sponsored by ISS and activated in 11 clinical sites in Italy in HIV-infected HAART-treated subjects (Ensoli F, Retrovirology 2015).In this study, subjects are randomized into two arms to receive 3 or 5 vaccinations monthly; each arm is composed of two treatment groups, receiving 7, 5 or 30 µg of Tat, respectively.Results obtained in 168 individuals after trial completion (48 weeks), as well as after a follow-up of 144 weeks for a subgroup of vaccines, indicated that Tat vaccination is safe, immunogenic and capable of reducing the immune dysregulation which persists despite HAART in treated individuals (Ensoli et al,PLoS ONE 2010). Anti-Tat Abs were induced in most patients (79%), with the highest frequency and durability in the Tat 30 µg groups (89%) particularly when given 3 times (92%) (Ensoli B.,PLoS ONE 2010; Ensoli F., Retrovirology 2015). Moreover, vaccination promoted a durable and significant restoration of T, B, natural killer (NK) cells, and CD4+ and CD8+ central memory subsets. Moreover, a significant reduction of blood proviral DNA was seen after week 72, particularly under PI-based regimens and with Tat 30 µg given 3 times (30 μg, 3x), reaching a predicted 70% decay after 3 years from vaccination with a half-life of 88 weeks. This decay was significantly associated with anti-Tat IgM and IgG Abs and neutralization of Tat-mediated entry of oligomeric Env in dendritic cells, which predicted HIV-1 DNA decay. Finally, the 30 μg, 3x group was the only one showing significant increases of NK cells and CD38+HLA-DR+/CD8+ T cells, a phenotype associated with increased killing activity in elite controllers (Ensoli F., Retrovirology 2015). These data indicate that Tat immunization represents a promising pathogenesis-driven intervention to intensify HAART efficacy (Ensoli et al,PLoS ONE 2010).

DETAILED DESCRIPTION:
Based on this, the ISS T-003 study in South Africa was started; the study was a phase II, randomized, double-blinded, placebo controlled, clinical trial to evaluate the immunogenicity (as a primary end-point) and the safety (as a secondary end-point), of a therapeutic, recombinant, biologically active HIV-1 Tat vaccine in HIV-1 infected, anti-Tat antibody negative, ARV-treated adult volunteers with chronically suppressed HIV-1 infection as indicated by a HIV-1 plasma viraemia < 400 copies/ml, and a CD4+ T cell count ≥ 200 cells/μl, at screening and documented at least once during the 12 month period prior to screening, irrespective of the pre-ARV CD4 nadir.

After a screening period of up to 21 days, the study duration will be 48 weeks, including an 8 week treatment phase (during which 3 vaccinations will be administered at 4-week intervals) and a 40 week follow-up phase.

This study will be conducted at 1 clinical site in South Africa. 200 Subjects were randomized in a 1:1 ratio to one of the two treatment groups (Tat 30 mcg or placebo administered intradermally, 3 times).

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers aged 18-45 years (inclusive)
* Anti-Tat antibody negative
* HIV-1 infected individuals currently receiving treatment with ARVs
* Chronically suppressed HIV-1 infection as indicated by a HIV-1 plasma viraemia < 400 copies/ml and a CD4+ T cell count ≥ 200 cells/μl at screening, and documented at least once during the 12 month period prior to screening, irrespective of the pre-ARV CD4 nadir.
* Negative pregnancy test for females of childbearing potential (not sterilized and still menstruating or within 1 year of the last menses) to be performed during the screening phase and immediately before each vaccination, and use of an acceptable method of contraception (double barrier methods, combined oral contraceptives, injectable contraceptives or intra-uterine devices) for at least 3 weeks prior to the first vaccination and for the duration of the study
* Has provided written informed consent.
* Agrees to stay in contact with the research site for the duration of the study

Exclusion Criteria:

* Acute illness on Study Day 0
* Body temperature >=37.5 °C on Study Day 0
* Any current AIDS-related opportunistic disease
* Any current neoplastic disease
* Known history of malignant neoplastic diseases [NOTE: Subjects with known history of non-malignant neoplastic diseases that are completely resolved according to the fulfilment of all the specific recovery criteria, in agreement with the current guidelines in medical oncology, are eligible]
* Known history of encephalopathy, neuropathy or unstable CNS pathology, immunodeficiency, autoimmune disease, angina or cardiac arrhythmias, or any other clinically significant medical problems in the opinion of the investigator
* Any evidence, as judged by the investigator, of unstable cardio-vascular disease (e.g. unstable hypertensive disease needing modification or introduction of an anti-hypertensive treatment)
* Chest radiography showing evidence of active or acute cardiac or pulmonary disease within 6 months prior to the study screening visit [Note if no previous chest X-ray available, this will be performed at screening];
* Known history of anaphylaxis or serious adverse reactions to vaccines
* Known history of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g. Steven-Johnson syndrome, bronchospasm, or hypotension)
* Active pulmonary tuberculosis within 12 months of screening as evidenced by chest radiography and/or medical history.
* Any known medical or psychiatric condition which precludes subject compliance with the protocol, specifically, persons with psychotic disorders, major affective disorders and/or suicidal ideation are to be excluded
* Current use of psychotropic drugs prescribed for major psychotic disorders
* Concomitant participation in any study with an investigational product or device
* Current or prior therapy with immunomodulator, immunosuppressive and/or anticoagulant drugs within 30 days prior to administration of the investigational product
* Live attenuated vaccines within 60 days of the first administration of the investigational product [NOTE: Medically indicated sub-unit or killed vaccines (e.g., influenza, pneumococcal, hepatitis A and B) are permitted, but must have been administered at least 4 weeks prior to the first administration of the investigational product]
* Known receipt of blood products or immunoglobulins during the year prior to screening
* Previous participation in an HIV-1 vaccine trial (subjects who are known to have previously participated in the placebo arm of an HIV-1 vaccine trial, and so have never received an investigational HIV-1 vaccine, are eligible for inclusion)
* Known drug and/or alcohol abuse in the year prior to screening
* Use in the last 6 months or concomitant use of anti-CCR5 inhibitors and/or integrase inhibitors and/or fusion inhibitors
* Pregnant or lactating females

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of Tat protein | up to 48 weeks
  Induction of specific anti-Tat humoral immune response in terms of IgM, IgG or IgA anti-Tat antibodies.
  The induction, magnitude and persistence of the humoral response to the administered vaccination schedule will be compared between the active and placebo groups.

SECONDARY OUTCOMES:
safety of the Tat protein | baseline; up to 48 weeks
  Changes in physical examination findings from baseline;
safety of the Tat protein | baseline; up to 48 weeks
  Changes in vital signs from baseline;
safety of the Tat protein | up to 48 weeks
  Adverse events (including local and systemic reactions to the vaccination schedule occurring during the course of the study);
safety of the Tat protein | baseline; up to 48 weeks
  Changes in standard laboratory safety parameters from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Barbara BE Ensoli, MD, Study Director — Istituto Superiore Sanita
Locations (1):
- Medunsa Clinical Research Unit (MeCRU), Medunsa, Gaueg, South Africa

REFERENCES:
- [Background] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Tripiciano A, Longo O, Bellino S, Francavilla V, Paniccia G, Arancio A, Scoglio A, Collacchi B, Ruiz Alvarez MJ, Tambussi G, Tassan Din C, Palamara G, Latini A, Antinori A, D'Offizi G, Giuliani M, Giulianelli M, Carta M, Monini P, Magnani M, Garaci E. The preventive phase I trial with the HIV-1 Tat-based vaccine. Vaccine. 2009 Dec 11;28(2):371-8. doi: 10.1016/j.vaccine.2009.10.038. Epub 2009 Oct 29. PMID 19879233
- [Background] Longo O, Tripiciano A, Fiorelli V, Bellino S, Scoglio A, Collacchi B, Alvarez MJ, Francavilla V, Arancio A, Paniccia G, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Phase I therapeutic trial of the HIV-1 Tat protein and long term follow-up. Vaccine. 2009 May 26;27(25-26):3306-12. doi: 10.1016/j.vaccine.2009.01.090. Epub 2009 Feb 7. PMID 19208456
- [Background] Ensoli B, Bellino S, Tripiciano A, Longo O, Francavilla V, Marcotullio S, Cafaro A, Picconi O, Paniccia G, Scoglio A, Arancio A, Ariola C, Ruiz Alvarez MJ, Campagna M, Scaramuzzi D, Iori C, Esposito R, Mussini C, Ghinelli F, Sighinolfi L, Palamara G, Latini A, Angarano G, Ladisa N, Soscia F, Mercurio VS, Lazzarin A, Tambussi G, Visintini R, Mazzotta F, Di Pietro M, Galli M, Rusconi S, Carosi G, Torti C, Di Perri G, Bonora S, Ensoli F, Garaci E. Therapeutic immunization with HIV-1 Tat reduces immune activation and loss of regulatory T-cells and improves immune function in subjects on HAART. PLoS One. 2010 Nov 11;5(11):e13540. doi: 10.1371/journal.pone.0013540. PMID 21085635
- [Background] Bellino S, Francavilla V, Longo O, Tripiciano A, Paniccia G, Arancio A, Fiorelli V, Scoglio A, Collacchi B, Campagna M, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Parallel conduction of the phase I preventive and therapeutic trials based on the Tat vaccine candidate. Rev Recent Clin Trials. 2009 Sep;4(3):195-204. doi: 10.2174/157488709789957529. PMID 20028332
- [Background] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Monini P, Magnani M, Garaci E. The therapeutic phase I trial of the recombinant native HIV-1 Tat protein. AIDS. 2008 Oct 18;22(16):2207-9. doi: 10.1097/QAD.0b013e32831392d4. PMID 18832884
- [Background] Ensoli B, Fiorelli V, Ensoli F, Cafaro A, Titti F, Butto S, Monini P, Magnani M, Caputo A, Garaci E. Candidate HIV-1 Tat vaccine development: from basic science to clinical trials. AIDS. 2006 Nov 28;20(18):2245-61. doi: 10.1097/QAD.0b013e3280112cd1. No abstract available. PMID 17117011
- [Background] Butto S, Fiorelli V, Tripiciano A, Ruiz-Alvarez MJ, Scoglio A, Ensoli F, Ciccozzi M, Collacchi B, Sabbatucci M, Cafaro A, Guzman CA, Borsetti A, Caputo A, Vardas E, Colvin M, Lukwiya M, Rezza G, Ensoli B; Tat Multicentric Study Group. Sequence conservation and antibody cross-recognition of clade B human immunodeficiency virus (HIV) type 1 Tat protein in HIV-1-infected Italians, Ugandans, and South Africans. J Infect Dis. 2003 Oct 15;188(8):1171-80. doi: 10.1086/378412. Epub 2003 Sep 30. PMID 14551888
- [Background] Rezza G, Fiorelli V, Dorrucci M, Ciccozzi M, Tripiciano A, Scoglio A, Collacchi B, Ruiz-Alvarez M, Giannetto C, Caputo A, Tomasoni L, Castelli F, Sciandra M, Sinicco A, Ensoli F, Butto S, Ensoli B. The presence of anti-Tat antibodies is predictive of long-term nonprogression to AIDS or severe immunodeficiency: findings in a cohort of HIV-1 seroconverters. J Infect Dis. 2005 Apr 15;191(8):1321-4. doi: 10.1086/428909. Epub 2005 Mar 14. PMID 15776379
- [Background] Bellino S, Tripiciano A, Picconi O, Francavilla V, Longo O, Sgadari C, Paniccia G, Arancio A, Angarano G, Ladisa N, Lazzarin A, Tambussi G, Nozza S, Torti C, Foca E, Palamara G, Latini A, Sighinolfi L, Mazzotta F, Di Pietro M, Di Perri G, Bonora S, Mercurio VS, Mussini C, Gori A, Galli M, Monini P, Cafaro A, Ensoli F, Ensoli B. The presence of anti-Tat antibodies in HIV-infected individuals is associated with containment of CD4+ T-cell decay and viral load, and with delay of disease progression: results of a 3-year cohort study. Retrovirology. 2014 Jun 24;11:49. doi: 10.1186/1742-4690-11-49. PMID 24961156
- [Background] Monini P, Cafaro A, Srivastava IK, Moretti S, Sharma VA, Andreini C, Chiozzini C, Ferrantelli F, Cossut MR, Tripiciano A, Nappi F, Longo O, Bellino S, Picconi O, Fanales-Belasio E, Borsetti A, Toschi E, Schiavoni I, Bacigalupo I, Kan E, Sernicola L, Maggiorella MT, Montin K, Porcu M, Leone P, Leone P, Collacchi B, Palladino C, Ridolfi B, Falchi M, Macchia I, Ulmer JB, Butto S, Sgadari C, Magnani M, Federico MP, Titti F, Banci L, Dallocchio F, Rappuoli R, Ensoli F, Barnett SW, Garaci E, Ensoli B. HIV-1 tat promotes integrin-mediated HIV transmission to dendritic cells by binding Env spikes and competes neutralization by anti-HIV antibodies. PLoS One. 2012;7(11):e48781. doi: 10.1371/journal.pone.0048781. Epub 2012 Nov 13. PMID 23152803
- [Background] Ensoli B, Cafaro A, Monini P, Marcotullio S, Ensoli F. Challenges in HIV Vaccine Research for Treatment and Prevention. Front Immunol. 2014 Sep 8;5:417. doi: 10.3389/fimmu.2014.00417. eCollection 2014. PMID 25250026
- [Background] Ensoli F, Cafaro A, Casabianca A, Tripiciano A, Bellino S, Longo O, Francavilla V, Picconi O, Sgadari C, Moretti S, Cossut MR, Arancio A, Orlandi C, Sernicola L, Maggiorella MT, Paniccia G, Mussini C, Lazzarin A, Sighinolfi L, Palamara G, Gori A, Angarano G, Di Pietro M, Galli M, Mercurio VS, Castelli F, Di Perri G, Monini P, Magnani M, Garaci E, Ensoli B. HIV-1 Tat immunization restores immune homeostasis and attacks the HAART-resistant blood HIV DNA: results of a randomized phase II exploratory clinical trial. Retrovirology. 2015 Apr 29;12:33. doi: 10.1186/s12977-015-0151-y. PMID 25924841
- [Background] Cafaro A, Tripiciano A, Sgadari C, Bellino S, Picconi O, Longo O, Francavilla V, Butto S, Titti F, Monini P, Ensoli F, Ensoli B. Development of a novel AIDS vaccine: the HIV-1 transactivator of transcription protein vaccine. Expert Opin Biol Ther. 2015;15 Suppl 1:S13-29. doi: 10.1517/14712598.2015.1021328. Epub 2015 Jun 22. PMID 26096836
- [Derived] Ensoli B, Nchabeleng M, Ensoli F, Tripiciano A, Bellino S, Picconi O, Sgadari C, Longo O, Tavoschi L, Joffe D, Cafaro A, Francavilla V, Moretti S, Pavone Cossut MR, Collacchi B, Arancio A, Paniccia G, Casabianca A, Magnani M, Butto S, Levendal E, Ndimande JV, Asia B, Pillay Y, Garaci E, Monini P; SMU-MeCRU study group. HIV-Tat immunization induces cross-clade neutralizing antibodies and CD4(+) T cell increases in antiretroviral-treated South African volunteers: a randomized phase II clinical trial. Retrovirology. 2016 Jun 9;13(1):34. doi: 10.1186/s12977-016-0261-1. PMID 27277839
- See also: Related info — http://www.hiv1tat-vaccines.info